CLINICAL TRIAL: NCT02916706
Title: Efficacy and Safety of Teneligliptin in Chinese Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-513-C02
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Results first posted 2022-01-28 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Teneligliptin 20mg (Experimental): Teneligliptin (20mg once daily) for 24 weeks
  Interventions: Drug: Teneligliptin 20mg
- Placebo (Placebo Comparator): Placebo for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teneligliptin 20mg
  Arms: Teneligliptin 20mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is designed as a prospective, multi-centre, parallel group, double-blind randomized, placebo-controlled, phase 3 clinical study to evaluate the efficacy and safety of MP-513 (Teneligliptin).

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent form has been obtained from the subject, in accordance with International Conference on Harmonisation guidelines on Good Clinical Practice (ICH GCP), before any screening or study related procedures take place.
* The subject is aged ≥18 years at signature of the informed consent form.
* Hospitalization status: outpatient.
* The subject has had a documented diagnosis of type 2 diabetes mellitus for at least 3 months at the screening visit (Day -28).
* The subject is undergoing diet and exercise therapy, and diet and exercise regimen has not been changed for at least 8 consecutive weeks at the screening visit (Day -28). Subjects who cannot do exercise due to complication are not limited to this criteria.
* The subject's glycosylated fraction of haemoglobin(HbA1c) is ≥ 7.0% and < 10.0% at the screening visit (Day -28) and on Day -14.

Exclusion Criteria:

* The subject has a history of type 1 diabetes mellitus or a secondary form of diabetes.
* The subject has received insulin within 1 year prior to the screening visit (Day -28), with the exception of insulin therapy during hospitalization or insulin therapy for medical conditions not requiring hospitalization (< 2 weeks' duration).
* The subject has received an anti-diabetic drug within 8 weeks prior to the screening visit (Day -28).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2016-09; Primary Completion 2018-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational center, Beijing, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Teneligliptin 20mg | Placebo
Started | 127 | 127
FAS | 125 | 126
Completed | 112 | 96
Not Completed | 15 | 31
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Other | 5 | 19

BASELINE CHARACTERISTICS:
Population: FAS: All subjects in the randomized set who have received at least one dose of study medication during the double-blind treatment period and have at least one post-baseline efficacy observation. Subjects who were not diagnosed with type 2 diabetes mellitus were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Teneligliptin 20mg | Placebo | Total
Number analyzed (Participants) | 125 | 126 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (10.2) | 56.0 (10.2) | 54.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 47 | 87
  Male | 85 | 79 | 164
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 125 | 126 | 251
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 24
Description: The change in HbA1c from baseline to Week 24 in Teneligliptin compared to Placebo was performed on FAS.
Time Frame: at Day 1(baseline) and Week 24
Population: All subjects in the randomized set who have received at least one dose of study medication during the double-blind treatment period and have at least one post-baseline efficacy observation. Subjects who were not diagnosed with type 2 diabetes mellitus were excluded.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Teneligliptin 20mg | Placebo
Number analyzed (Participants) | 125 | 126
percentage of HbA1c | -0.95 (0.06) | -0.14 (0.06)

2. Secondary Outcome: The Changes in Fasting Plasma Glucose (FPG) at Week 24
Description: The change in FPG from baseline to Week 24 in Teneligliptin compared to Placebo was performed on FAS.
Time Frame: at Day 1(baseline) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Teneligliptin 20mg | Placebo
Number analyzed (Participants) | 125 | 126
mg/dL | -21.9 (2.5) | -1.4 (2.5)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Teneligliptin 20mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/127
Serious Adverse Events (participants affected / at risk) | 6/127 | 4/127
Other Adverse Events (participants affected / at risk) | 69/127 | 50/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teneligliptin 20mg (N=127) | Placebo (N=127)
Angina pectoris (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Teneligliptin 20mg (N=127) | Placebo (N=127)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 6
Hepatic function abnormal (Hepatobiliary disorders) | 7 | 2
Upper respiratory tract infection (Infections and infestations) | 30 | 20
Protein urine present (Investigations) | 7 | 5
Urine ketone body present (Investigations) | 9 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 | 9
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 7
Proteinuria (Renal and urinary disorders) | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-04-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT02916706/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT02916706/SAP_001.pdf